CLINICAL TRIAL: NCT00181363
Title: Mamma Board Project: Prone Breast Irradiation for Pendulous Breasts
Brief Title: Prone Breast Irradiation for Pendulous Breasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03.1446L
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast conserving surgery; Radiotherapy; Pendulous breasts
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mamma board (Experimental): use of the mamma board during radiotherapy
  Interventions: Device: Mamma board

INTERVENTIONS:
Device: Mamma board — use of mamma board during radiotherapy
  Other Names: radiation, prone breast, mammaboard

SUMMARY:
We hypothesize that for large pendulous breasts, breast irradiation in supine and prone position are equivalent with regard to coverage of the PTV, but with a better dose homogeneity in prone position and a smaller radiation exposure of lung and heart.The purpose of this study is to compare the 3-D dose distribution in PTV(Planning Target Volume) and normal tissues in prone position versus supine position.

DETAILED DESCRIPTION:
Local excision followed by adjuvant radiotherapy has become standard treatment for women with early-stage breast cancer. Adjuvant radiotherapy may encounter technical difficulties in patients with pendulous breasts when treated in supine position.

Based upon literature and our own preliminary experiences, we hypothesize that for large pendulous breasts, breast irradiation in supine and prone position are equivalent with regard to coverage of the PTV, but with a better dose homogeneity in prone position and a smaller radiation exposure of lung and heart. However, no quantitative data are yet available to test this hypothesis. Therefore, the aim of our study is to compare the 3-D dose distribution in PTV and normal tissues in prone position versus supine position. For treatment in prone-position an in-house developed device, the "mammaboard" was used.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have had breast-conserving surgery for breast cancer or DCIS (Ductal Carcinoma in Situ)
* No indication for radiotherapy of regional nodes
* Large, pendulous breasts (bra size D and over)

Exclusion Criteria:

* Regional radiotherapy is indicated
* Unable to lie in prone position

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-12; Primary Completion 2006-07 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Buijsen, MD, Principal Investigator — Maastricht Radiation Oncology
Locations (1):
- Maastricht Radiation Oncology, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mamma Board: Mamma board used during radiotherapy
Period: Overall Study
Arm/Group | Mamma Board
Started | 10 (10)
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Mamma board
Arm/Group | Group 1
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 10

OUTCOME MEASURES:

1. Primary Outcome: Dose Homogeneity 1: PTV
Description: Quantitatively compare the 3 D dose distribution in the PTV (Planning Target Volume) and normal tissues in prone position versus supine position
Time Frame: 1 day after treatment planning
Population: To investigate dose homogeneity and maximum doses, Dmin (minimum Dose), Dmax (maximum Dose) and Dmean (mean Dose) were calculated for prone position versus supine position.
Measure: Mean (Standard Deviation); unit: Gy
Groups:
- Prone: Prone position
- Supine: Supine position
Arm/Group | Prone | Supine
Number analyzed (Participants) | 10 | 10
Gy
  Dmin (Gy) PTV | 9.8 (6.7) | 8.2 (5.6)
  Dmean (Gy) PTV | 48.2 (1.2) | 49.8 (0.8)
  Dmax (Gy) PTV | 53.6 (0.6) | 54.8 (1.4)
Statistical Analysis 1: Comparison: Prone vs Supine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Dose Homogeneity 2: V105% and V107%
Description: Quantitatively compare the 3 D dose distribution in the PTV (Planning Target Volume) in prone position versus supine position
Time Frame: 1 day after treatment planning
Population: To investigate dose homogeneity V105% (volume of tissue receiving more than 105% of the prescribed dose) and V107% (volume of tissue receiving more than 107% of the prescribed dose) were calculated for prone position versus supine position.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Prone | Supine
Number analyzed (Participants) | 10 | 10
cc
  V105% PTV | 1.5 (1.2) | 9.1 (9.9)
  V107% PTV | 0.1 (0.3) | 2.8 (4.8)
Statistical Analysis 1: Comparison: Prone vs Supine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: PTV Coverage in Organs at Risk: MLD (Gy)
Description: Doses in organs at risk: lung MLD (Mean Lung Dose)
Time Frame: during treatment planning
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Prone | Supine
Number analyzed (Participants) | 10 | 10
Gy | 0.9 (0.6) | 4.1 (1.6)
Statistical Analysis 1: Comparison: Prone; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: PTV Coverage in Organs at Risk: Heart V30
Description: Doses in organs at risk: heart V30: the volumes (%) of the heart that received >= 30Gy
Time Frame: during treatment planning
Measure: Mean (Standard Deviation); unit: percentage of V30
Arm/Group | Prone | Supine
Number analyzed (Participants) | 10 | 10
percentage of V30 | 2.4 (3.0) | 7.3 (4.6)
Statistical Analysis 1: Comparison: Prone vs Supine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Dose Homogeneity 3: V95 %
Description: PTV coverage (% of PTV < 95% of prescribed dose) in prone position versus supine position
Time Frame: 1 day after treatment planning
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Prone | Supine
Number analyzed (Participants) | 10 | 10
cc
  V95%PTV | 78.6 (5.6) | 91.4 (4.1)
  V95%CTV | 85.0 (4.2) | 93.3 (4.0)
Statistical Analysis 1: Comparison: Prone vs Supine; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: during treatment
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes